CLINICAL TRIAL: NCT02439047
Title: Non-stick Patch of Mesothelial Cells in a Hydrogel Matrix : Exploratory Analysis Assessing the Morphotype and Mesothelial Phenotype After Culture From 2 Cells Sources of Human Origin.
Brief Title: Preliminary Study to the Manufacturing of a Non-stick Membrane for Surgery Using Patient's Own Cells (MESO-PATCH)
Acronym: MESO-PATCH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty of carrying out the analysis and low recruitment
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MESO-PATCH-1408
Record Dates: First submitted 2015-04-23; First posted 2015-05-08 (Estimated); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Cancer
Keywords: reconstructive surgery; abdominal surgery
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Biological samples collection (Experimental): -Peritoneal samples : will be collected during abdominal surgery
  A biopsy from 1 to 2 cm2 will be performed in healthy peritoneum
  -Adipose tissue samples : will be collected during surgery for breast reconstruction
  Interventions: Procedure: Biological samples collection

INTERVENTIONS:
Procedure: Biological samples collection — -Peritoneal samples : will be collected during abdominal surgery
  A biopsy from 1 to 2 cm2 will be performed in healthy peritoneum
  - Adipose tissue samples : will be collected during surgery for breast reconstruction

SUMMARY:
The objective of this study, which will be realised in vitro on human samples, is to test 2 cell sources isolated from peritoneum for adult mesothelial cells (peritoneal samples) and from adipose tissue for the adipose stem cells (adipose tissue samples). The latter will be differentiated towards the mesothelial phenotype and morphotype. The 2 routes will be compared and the most satisfactory one will be chosen to make a non-stick patch.

DETAILED DESCRIPTION:
* Patient information and collection of a signed informed consent
* Clinical data collection: surgery date, age, weight, height, medical and surgical history
* Prospective collection of peritoneal and adipose biopsies of patients during their surgery at the Oscar Lambret Center (Dr L. BRESSON)
* Transportation of the samples to the 1008 INSERM Unit.
* Isolation of cells from the samples : mesothelial cells from the peritoneum and adipose stem cells from adipose tissue
* Cell culture and expansion of mesothelial cells; and cell culture and differentiation of adipose stem cells
* Identification by the morphotype and phenotype of mesothelial cells
* Comparison of the results according to the cell source, peritoneum or adipocyte, to the purity of cells and to the efficacy of the expansion

ELIGIBILITY:
Inclusion Criteria:

* Aged more than 18 years old,
* Planned surgery For peritoneal samples : abdominal surgery (laparotomy or coelioscopy) For adipose tissue samples : breast reconstructive surgery (lipomodelage)
* Informed and signed consent

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Patient under guardianship or tutorship
* For peritoneal samples : previous abdomino-pelvic radiotherapy or abdominal surgery ; peritoneal carcinosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-06; Primary Completion 2015-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Morphotype/Phenotype expression | 1 year
  Mesothelial morphotype and phenotype expression of the 2 types of cells after culture

CONTACTS AND LOCATIONS:
Overall Officials: Lucie BRESSON, MD, Principal Investigator — Centre Oscar Lambret; Feng Chai, MD, Study Director — INSERM U1008
Locations (1):
- Centre Oscar Lambret, Lille, France

IPD SHARING:
Plan to Share IPD: No